CLINICAL TRIAL: NCT02391272
Title: A Multicenter Open-labeled Pilot Study on Recombinant Human Thrombopoietin in Management of Immune Thrombocytopenia in Pregnancy
Brief Title: A Multicenter Study on Recombinant Human Thrombopoietin in Management of ITP in Pregnancy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shandong University (Other)
Collaborators: The Affiliated Hospital of Qingdao University (Other); The Second Hospital of Hebei Medical University (Other); Institute of Hematology & Blood Diseases Hospital, China (Other); Southern Medical University, China (Other)
Responsible Party: Principal Investigator, Ming Hou, Professor and Director, Shandong University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ITP-pregnancy-rhTPO-Multi
Record Dates: First submitted 2015-03-02; First posted 2015-03-18 (Estimated); Last update posted 2020-03-20 (Actual); Status verified 2016-03

CONDITIONS: Immune Thrombocytopenia; Pregnancy
Keywords: recombinant human thrombopoietin; immune thrombocytopenia; pregnancy
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- rhTPO (Experimental): rhTPO will be given intravenously at a dose of 300U/kg every day. Dose will be tapered to 300U/kg every other day when platelet count rise over 50×10^9/L. Maintenance will be continued after delivery and the dose will be further reduced to 300U/kg per week.
  Interventions: Drug: rhTPO

INTERVENTIONS:
Drug: rhTPO
  Other Names: TPIAO

SUMMARY:
The project was undertaking by Qilu Hospital of Shandong University and other well-known hospitals in China. Aims at evaluating efficacy and safety of rhTPO in management of ITP in pregnancy.

DETAILED DESCRIPTION:
The investigators are undertaking a multicenter, open-labeled, pilot study of 30 ITP patients in pregnancy from Qilu Hospital of Shandong University and other well-known hospitals in China. ITP patients in pregnancy who failed to respond to prednisone, IVIG and developed refractoriness to platelet transfusion will be given rhTPO intravenously at a dose of 300U/kg every day. Dose will be tapered to 300U/kg every other day when platelet count rise over 50×10^9/L. Maintenance will be continued after delivery and the dose will be further reduced to 300U/kg per week. Platelet count, bleeding and other symptoms will be evaluated before and after treatment. Adverse events will be recorded throughout the study.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is between 18-50 years old.
2. After 12 weeks gestation.
3. Diagnosed with ITP meeting the diagnostic criteria for immune thrombocytopenia.
4. Patients who have no response or relapsed after Corticosteroid or IVIG.
5. Patients developed refractoriness to platelet transfusion.
6. To show a platelet count < 30×10^9/L, and with bleeding manifestations.
7. Willing and able to sign written informed consent.

Exclusion Criteria:

1. Received chemotherapy or anticoagulants or other drugs affecting the platelet counts within 3 months before the screening visit.
2. Received second-line ITP-specific treatments (eg, cyclophosphamide, 6-mercaptopurine, vincristine, vinblastine, etc) within 3 months before the screening visit.
3. Current HIV infection or hepatitis B virus or hepatitis C virus infections.
4. Severe medical condition (lung, hepatic or renal disorder) other than chronic ITP. Unstable or uncontrolled disease or condition related to or impacting cardiac function (e.g., unstable angina, congestive heart failure, uncontrolled hypertension or cardiac arrhythmia)
5. Have a known diagnosis of other autoimmune diseases, established in the medical history and laboratory findings with positive results for the determination of antinuclear antibodies, anti-cardiolipin antibodies, lupus anticoagulant or direct Coombs test.
6. Patients who are deemed unsuitable for the study by the investigator.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2015-03; Primary Completion 2015-11 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Early response 1- Response rate (CR+R) | 7th day
  Response rate (CR+R) at the 7th day. CR is defined as platelet count ≥ 100×10^9/L, and R is defined as platelet count of >30×10^9/L with at least a doubling of the baseline value.
Early response 2- Response rate (CR+R) | 14th day
  Response rate (CR+R) at the 14th day.
Long-time response 1 (Platelet count) | 10th week
  Platelet count at 10th week.
Long-time response 2 (Platelet count) | 40 weeks' gestation
  Platelet count at 40 weeks' gestation.
Long-time response 3 (Platelet count) | one month after delivery
  Platelet count one month after delivery.
Safety (Adverse events) | 6 months after delivery
  Adverse events in patients and infants.

CONTACTS AND LOCATIONS:
Overall Officials: Ming Hou, MD PhD, Principal Investigator — Shandong University Qilu Hospital
Locations (1):
- Qilu Hospital, Shandong University, Jinan, Shandong, China

REFERENCES:
- [Derived] Kong Z, Qin P, Xiao S, Zhou H, Li H, Yang R, Liu X, Luo J, Li Z, Ji G, Cui Z, Bai Y, Wu Y, Shao L, Peng J, Ma J, Hou M. A novel recombinant human thrombopoietin therapy for the management of immune thrombocytopenia in pregnancy. Blood. 2017 Aug 31;130(9):1097-1103. doi: 10.1182/blood-2017-01-761262. Epub 2017 Jun 19. PMID 28630121